**Official Title:** RECOVER-SLEEP: A Platform Protocol for Evaluation of Interventions for Sleep Disturbances in Post-Acute Sequelae of SARS-CoV-2 Infection (PASC)

**NCT:** NCT06404086

IRB Document Date: 8 February 2024

Duke Clinical Research Institute (DCRI) / Protocol Number Pro00112484 / RECOVER-SLEEP


# MASTER INFORMED CONSENT FORM AND AUTHORIZATION TO USE AND DISCLOSE PROTECTED HEALTH INFORMATION

Sponsor / Study Title: Duke Clinical Research Institute (DCRI) / "RECOVER-SLEEP: A

Platform Protocol for Evaluation of Interventions for Sleep Disturbances in Post-Acute Sequelae of SARS-CoV-2 Infection

(PASC)"

\_Protocol Number: Pro00112484 / RECOVER-SLEEP

**Principal Investigator:** 

«PiFullName»

(Study Doctor)

Telephone: «IcfPhoneNumber»

Address: «PiLocations»

#### **Concise Summary**

This is a research study to find out if certain study interventions can help treat sleep disturbances that started or got worse following a COVID infection and have lasted for at least 12 weeks. Sleep disturbances include excessive drowsiness, problems falling and staying asleep, and problems with sleep-wake patterns. These sleep disturbances are known to be associated with Post-Acute Sequelae of SARS-CoV-2 Infection (PASC) or Long COVID. This study will look at the effects the study interventions may have on your ability to get better and recover from the sleep disturbances associated with Long COVID.

This study will enroll adults who experience sleep disturbances as a symptom of Long COVID and who have not had another COVID infection in the past 4 weeks. These studies are being supported by the National Institutes of Health (NIH) through the Researching COVID to Enhance Recovery (RECOVER) Initiative.

By signing this consent and authorization form, you are giving the study team permission to determine if one of our sleep research studies might be a good fit for your based upon your sleep symptoms. This Master Consent form covers the following study activities:

• **Screening:** You will be asked questions about your sleep symptoms. This allows the study team to determine how your symptoms have been affecting your daily life. If it appears



Duke Clinical Research Institute (DCRI) / Protocol Number Pro00112484 / RECOVER-SLEEP


that you are a good fit for one of the sleep studies, you will be screened for symptoms of obstructive sleep apnea. You will be asked about any evaluation or treatment you may have received for sleep apnea. If you have not been evaluated for sleep apnea in the past, or if you may have an untreated sleep apnea, you may be asked to complete homebased sleep apnea testing (HSAT) before participating in the study.

• **Sub-Study Assignment:** Once you have been evaluated for sleep-related breathing disorders, you will be screened for assignment to one of the active sleep sub-studies. This study has multiple sub-studies and they may be open to participant enrollment at the same time or at different times. Each sub-study contains 1 or more active study intervention group and an inactive study intervention group. An intervention could include a study drug, a study device, a behavioral approach, or a combination of these interventions.

You will be assigned to the sub-study that best matches the type of sleep disturbance you are experiencing. It is also possible that you will not qualify for any of the active sub-studies because your sleep symptoms are not severe enough. If your sleep symptoms qualify you for more than one active sub-study, you will be assigned to only one sub-study; you may participate in only one sub-study at a time.

Once assigned to the sub-study that best matches your symptoms, you will be asked to sign another consent and authorization form that covers specific details for that individual sub-study. Depending on the sub-study you are assigned, you will then be randomly assigned by chance (like rolling a die) to 1 or more study interventions, referred to as "randomization." Within each sub-study, you will have a chance of being assigned at random to either an active or inactive study intervention group. Each sub-study will include approximately 500 to 600 participants from many study sites across the United States. The number of participants in each sub-study will differ.

• **Sub-Study Description:** Your assigned sub-study consent will provide details regarding what study intervention(s) are included in your sub-study, how long you will be asked to participate in receiving the study intervention(s), and how long you will be asked to participate in the study.

If enrolled as a sub-study participant, you will be asked to do the following:

- Answer questions about your symptoms and quality of life
- Complete a Sleep Diary
- Wear an activity tracker (a Fitbit or similar device) to record your rest and activity patterns

Duke Clinical Research Institute (DCRI) / Protocol Number Pro00112484 / RECOVER-SLEEP


- Provide a blood sample
- Complete tests to measure your memory and thinking abilities (referred to as "brain quizzes")
- Complete various questionnaires

If you are involved in multiple RECOVER trials and/or the RECOVER longitudinal cohort, your study data (including a limited number of identifiers such as date of birth, dates of study and health events) may be linked between RECOVER studies and analyzed together across RECOVER studies.

There is no guarantee of benefit to you, and there are some possible risks from participating in this study. Possible risks, such as possible side effects and loss of confidentiality, are detailed later in this consent form. Every effort will be made to minimize these risks. You do not have to participate in this research to be treated for your condition. If you choose not to participate, your usual healthcare will not be affected.

#### STUDY CONSENT

You are being asked to participate in the study called "RECOVER-SLEEP: A Platform Protocol for Evaluation of Interventions for Sleep Disturbances in Post-Acute Sequelae of SARS-CoV-2 Infection (PASC)". "Sequelae" are conditions or symptoms that result from having a previous disease.

This study is part of the Researching COVID to Enhance Recovery (RECOVER) Initiative.

This study currently offers the following sub-studies:

- Hypersomnia (excessive daytime sleepiness)
- Complex PASC-Related Sleep Disturbances (CPSD) (trouble falling asleep, staying asleep, or sleeping at irregular times)

Your participation is voluntary. Please review the information in this consent form to help you decide if you want to take part in the study. The use of the study drug and some study devices in this study are investigational. An investigational use is one that is not approved by the United States Food and Drug Administration (FDA).

SD\_ICF\_V3.0\_ 

#### INTRODUCTION

#### Why am I being asked to take part in this study?

You are being asked to take part in this study because you are at least 18 years old, had a COVID infection that caused new or worsened nighttime sleep and/or daytime sleepiness, and have been experiencing worsened nighttime sleep and/or increased daytime sleepiness for at least 12 weeks since the COVID infection.

#### Why is this study being done?

The number of people experiencing Long COVID is increasing in both hospitals and communities, and the symptoms of Long COVID affect quality of life. This study aims to improve the quality of life for people with sleep-related Long COVID symptoms. This study will look at multiple study interventions and their ability to treat sleep disturbances associated with Long COVID. Results from this study may help researchers better understand the condition and how to treat it.

## **VOLUNTARY PARTICIPATION/POTENTIAL BENEFITS**

### What if I don't want to participate?

You do not have to participate if you do not want to. Participation is voluntary. If you decide not to participate, your usual healthcare will not be affected. If you decide to participate, you can stop at any time.



#### Will there be any benefit to others or me?

We do not know if you will benefit from taking part in this study. The study intervention(s) may have a role in treating sleep-related Long COVID symptoms. You may want to participate to help doctors learn how to best care for adults with Long COVID. The information learned from this study may benefit others like you in the future. If you have a home sleep apnea test (HSAT), you will be provided the results of this test, which can guide further evaluation and treatment. If indicated, based on results of testing, you may be provided with a positive airway pressure device (the most common medical treatment for sleep apnea). You may be given monitoring study devices for use during the study (for example, an activity tracker, like a Fitbit, and a portable blood pressure monitor). You may be able to keep these study devices for personal health monitoring after the study ends if these were provided to you.

#### Will I be told about any new findings?

Yes. You will learn of any new, important information that is discovered during the study and any information that may influence your decision to continue participating in the study.

SD\_ICF\_V3.0\_ 

#### WHAT YOU CAN EXPECT IF YOU DECIDE TO PARTICIPATE



#### How long will I be in this study?

The amount of time you are expected to participate in the research study will depend on which sub-study you are assigned. Participation in the current substudies may last between 13 and 15 weeks. This includes an end of study phone call about 4 weeks after the end of the study intervention. **Refer to your Sub-Study Consent for more information.** 

Your length of participation will depend on whether you need home sleep apnea testing (HSAT) prior to starting a study intervention. If you require testing and this reveals that you have moderate to severe obstructive sleep apnea, or another severe sleep-related breathing disorder, you will be asked to discuss the findings and possible need for treatment with your health care providers. The time needed to undergo this evaluation and possible treatment may take up to 6 weeks, after which you will be eligible to be re-evaluated to take part in this study, depending on your results and treatment compliance. If you do not require testing, it should take only a few days to find out whether a particular sub-study is a good fit for you.

## How will I be assigned to a Sub-Study?

The study team will ask you complete sleep screening questionnaires to assess which sub-study (for example, Hypersomnia or CPSD) would be best to address your symptoms. Based on your sleep screening test results, you will be assigned to a sub-study and you will be asked to sign another consent form specific to that sub-study. Within your sub-study, you will be randomized (like rolling a die) to at least one or more active or one placebo (inactive) study intervention(s).

#### Will I know to which study intervention (active or inactive) I have been assigned?

You will know which sub-study you are enrolled in. However, you, your study doctor, and the study team will not know if you are receiving the active or inactive intervention, but they can quickly find out for your safety or well-being.

#### Can I participate in this study if I am already enrolled in other studies?

It depends. As long as the other studies do not interfere with your eligibility for this study, such as taking certain medicine(s), you should be able to participate in this study. You should notify your study doctor if you are participating in any other studies.

#### Will other types of sleep disturbances and study interventions be studied later on?

Over time, this study may expand to test additional study interventions, including other study drugs, study devices, or behavioral study interventions, After the study is complete, researchers



Duke Clinical Research Institute (DCRI) / Protocol Number Pro00112484 / RECOVER-SLEEP


will analyze data from the studies to learn if the studied interventions affected participants' sleep health.

#### **SUB-STUDY INTERVENTIONS**

Information about the sub-study interventions, total length of participation, and number of inperson visits for each study are listed in the Sub-Study Consent Form.

If you decide to stop participating in the study before your study intervention has completed, you will be asked to come into the study site to complete activities (referenced in your Sub-Study Consent Form) so we can collect important study data.

#### **SCREENING**

Within 6 weeks of starting your study intervention(s), you will be asked several questions about your COVID symptoms, general health and well-being, and any new or worsening health problems you may have to make sure this study is a good fit for you. You may be able to answer these questions without coming into the study doctor's office. You will be asked to:

- Complete questionnaires about your current sleep symptoms and habits which take less than 15 minutes to complete
- Review your current medications
- Take a pregnancy test (urine or blood collection, at the study site's discretion), if you could become pregnant
- Give a nasal swab sample to test for COVID
- Answer questions about whether or not you have ever been diagnosed with a sleep related breathing disorder (SRBD) such as sleep apnea (see "Home Sleep Apnea Testing" below).

Home Sleep Apnea Testing (HSAT): As part of screening for sleep related breathing disorders, you will be asked if you have ever been diagnosed or treated for symptoms of sleep apnea. If you have been evaluated in the past for sleep apnea, you may be asked to provide permission to review your medical records to see what type of sleep apnea you have and how it was treated. If you have not been evaluated in the past, you may be asked to do home sleep apnea testing (HSAT) before being assigned to a sub-study. If that testing shows you have a high likelihood of having moderate or severe obstructive sleep apnea, you will be provided with the results and will be asked to discuss further testing and treatment with your study team. If treatment of sleep apnea with a positive airway pressure (PAP) device is recommended, the study can provide you with one of these devices (like a CPAP machine). At the end of the study, you may keep the PAP device that was provided. Once your sleep apnea is adequately treated



Duke Clinical Research Institute (DCRI) / Protocol Number Pro00112484 / RECOVER-SLEEP


and adherence to the treatment is verified, the study team will evaluate whether your sleep symptoms still qualify you for enrollment in a sub-study. If a HSAT shows that you have breathing problems during sleep but these problems are not related to obstructive sleep apnea, you will be asked to discuss further evaluation and treatment with your healthcare provider.

**Sub-Study Screening and Consent:** After the home sleep apnea testing (HSAT), if the study still appears to be a good match for you and you choose to participate, you will be asked to visit your study doctor's office for the sub-study screening (pre-randomization) visit. This visit may happen in one or more days, and some assessments may be able to be completed by phone and/or electronically, depending upon your needs. The purpose of this visit is to confirm your interest in participating and tell you about what to expect during the study.

#### You will be asked to:

- Repeat, if necessary, some activities referenced above
- Provide a blood sample for sub-study screening tests

Your study team will review your screening test results which will determine to which sub-study you should be assigned. Once assigned to a sub-study, you will be asked to sign the Sub-Study Consent Form. Additional sub-study activities will be referenced within that consent form.

#### **RANDOMIZATION**

This visit may happen over one or more days, and some assessments may be able to be completed by phone/ and/or electronically (internet-based), depending on your needs.

#### Once you have given consent to participate in a sub-study, you will undergo the following

- Repeat, if necessary, some activities from screening
- Be randomized (like rolling a die) to either an active study intervention group or an inactive study intervention group
- Receive your (blinded) study intervention(s)
- Have your height and weight measured
- Give a blood sample
- Review of home medications (only if the screening review was done more than 14 days prior)
- Receive a home stool collection kit with instructions
- Complete brain quizzes and various questionnaires (these all take less than 60 minutes to complete)
- Receive an activity tracker (a Fitbit or similar device) to record rest and activity patterns
  - These patterns are used to measure times when you are asleep and awake


- These study devices require the use of a compatible mobile device
  - If you do not have a mobile device or a data plan compatible with the activity tracker, then one may be provided. If a mobile device is provided, you may keep it at the end of the study.
- Receive instructions for an internet-based Sleep Diary (or receive a paper version, if needed) to record rest and activity patterns and factors that may influence sleep
  - These patterns are used to measure times when you are asleep and awake
- Report any new or worsening symptoms since screening

Refer to your Sub-Study Consent Form for additional activities.

#### **Personal Information**

If you decide to take part in the study, we will ask for your:

- Date of birth so we can confirm your age
- Social Security number so we can pay you for your time and complete the tax form
- Home address so we can send your payment to you
- Phone number and email address so we can contact you to see if you have any questions or problems during the study
- Contact information for a person you trust, like a family member or friend, so we can contact them if we cannot reach you. Your trusted contact may give us some information about your health if you are not able to



- Details about your COVID infection(s) and COVID vaccination status
- Your health history including sleep-specific history, general health, and well-being
- Your allergies and a list of medicines (prescription and non-prescription) you are taking

We will also ask you to sign a medical release form. This will allow the study team to access your medical record to review relevant health history and any hospitalizations that may occur while you are participating in the study.

#### **Blood Sample Collection**

We will ask you to give blood samples for study-specific tests and for biorepository storage 2 times during the study (as referenced in your Sub-Study Consent Form). We will take about 5 ½ tablespoons (80 ml) of blood from your arm each visit to run study-specific tests and to store samples for future research, if possible. See the "Biorepository: Research Use of Data and Biospecimens" section for more information.





SD\_ICF\_V3.0\_ 

### **Stool Sample Collection**

You will be given a stool sample home kit and instructions 2 times during the study (as referenced in your Sub-Study Consent Form). We will ask that you collect the stool and place it in the provided collection container during your next bowel movement. We will ask you to mail the stool sample per our instructions. The stool samples may be used for future research; see the "Biorepository: Research Use of Data and Biospecimens" section for more information.

#### **Sleep Apnea Treatment Information**

The condition being studied is obstructive sleep apnea, which is a sleep disorder, characterized by pauses in breathing during sleep. The treatment for this condition is a device that delivers positive air pressure (PAP) through a mask placed over your nose while you sleep.

As a participant in this study, there is a possibility that you may receive a PAP device called the AirSense 11 (ResMed). PAP device consists of an air pump that provides a continuous flow of air through a tube and a mask that covers your nose or both your nose and mouth. The device gently sends air through the mask to keep your airways open while you sleep. The device also warms and humidifies the air for better comfort.

The device will send your usage data to a secure online system called AirView. This lets your healthcare team monitor your progress and make sure the treatment is working effectively. All your data is kept private and secure.

It's important for you to know that the research team will be keeping an eye on how you're doing with the device. If they notice anything that suggests your treatment could be improved – like if the mask isn't fitting right, or if the device settings need adjusting – someone from the team might reach out to you.

Also, we encourage you to sign up for myAir, a user-friendly program on your phone or computer. It tracks your therapy, gives you daily scores, and offers tips and encouragement. This can help you see how well you're doing and learn ways to make your treatment even better.

SD\_ICF\_V3.0\_ 

#### WEEK 1

## During week 1, which occurs immediately following the week 0 visit, you will be asked to do the following:

- Use the activity tracker when you are awake and asleep
  - You will be asked to wear this study device for 7 days before starting your study intervention
- Complete the Sleep Diary
  - You will be asked to complete this Diary for 7 days before starting your study intervention

Refer to your Sub-Study Consent Form for additional sub-study-specific activities.

#### **WEEK 2 TO FINAL IN-PERSON VISIT**

Refer to your Sub-Study Consent Form for information about the total length of the study intervention(s) and any sub-study specific additional activities. The final in-person visit occurs at the same time as when you will stop the study intervention(s). During this time, you will be asked to:

- Use the activity tracker when you are awake and asleep
  - You will be encouraged to wear this study device for the duration of the substudy, but the use of this study device is optional during this time

**Sub-Study Titration Period:** Refer to your Sub-Study Consent Form regarding the study titration period, if applicable.

**Middle of Sub-Study Phone Call:** You will be asked to answer a phone call around the middle of this study. The timing of this call will depend on sub-study assignment and will be outlined in the Sub-Study Consent Form.

During this call, we will ask you to:

- Provide details about how you are completing your study interventions
- Report any new or worsening symptoms
- Review your current medications

If you report certain symptoms, you may be asked to make an additional in-person visit to your study site.

#### 7 days prior to your scheduled final in-person visit we will ask you to:

• Use the activity tracker when you are awake and asleep

Complete the Sleep Diary

### **END OF INTERVENTION (FINAL IN-PERSON VISIT)**

You will be asked to come to the study site for an in-person visit after your complete your study intervention(s). Refer to your Sub-Study Consent Form for information about the total length of the study intervention(s) and any sub-study specific additional activities.

## During this visit, which will mark the end of the intervention, you will be asked to do the following:

- Complete questionnaires about your current sleep habits (these take less than 10 minutes to complete)
- Review your current medications
- Have your weight measured
- Complete brain quizzes and various questionnaires (these all take less than 60 minutes to complete)
- Give a blood sample
- Receive a home stool collection kit with instructions
- Provide details about how you completed your study intervention(s)
- Report any new or worsening symptoms
- Return the remaining study drug and study devices, if applicable

Additionally, we will ask if any of the following information about your health has changed, including:

- Your health history including sleep-specific history, general health, and well-being
- Your allergies and the list of medicines (prescription and non-prescription)
   you are taking

If you decide to stop participating in the study before the study ends, you will be asked to come into the study site to complete a visit so we can collect important study data. This visit will include all of the activities referenced above for the Final Clinic Visit.

## **FINAL PHONE CALL (END OF STUDY)**

A study team member will call you about 4 weeks after you complete your final clinic visit.

#### 7 days prior to this scheduled call, we will ask you to:

Use the activity tracker when you are awake and asleep



 $SD\_ICF\_V3.0\_$ 

Duke Clinical Research Institute (DCRI) / Protocol Number Pro00112484 / RECOVER-SLEEP


## During this call, we will ask you to:

- Report any new or worsening symptoms
- Complete questionnaires (these take less than 10 minutes to complete)



Duke Clinical Research Institute (DCRI) / Protocol Number Pro00112484 / RECOVER-SLEEP


## STUDY AND SUB-STUDY SCHEDULE OF ACTIVITIES

| Screening ** | Randomization ** | Week 1 ** | Week 2 to Final In-Person Visit ** |
|---|---|---|---|
| Clinic Visit and At-Home Activities (Phone and Internet-Based) | Clinic Visit | At-Home Activities (Phone and Internet-Based) | At-Home Activities (Phone and Internet-<br>Based) |
| | *** | | |
| <ul> <li>Master Consent Form signing (this document)</li> <li>Sleep related breathing disorder screening, including home sleep apnea testing, if applicable</li> <li>Questionnaires</li> <li>Demographics</li> <li>Review medications</li> <li>Medical and sleep history</li> <li>Pregnancy test (urine or blood collection), if applicable</li> <li>Nasal swab</li> <li>Sub-Study Consent Form signing</li> <li>Blood collection for sub-study screening tests</li> </ul> | <ul> <li>Repeat any screening activities, as necessary</li> <li>Questionnaires and brain quizzes</li> <li>Blood collection</li> <li>Measure height and weight</li> <li>Stool Sample*</li> <li>Receive activity tracker (and other study devices, if applicable, as specified in your Sub-Study Consent Form)</li> <li>Receive the Sleep Diary</li> <li>Safety assessment</li> <li>Receive study intervention assignment and corresponding intervention(s)</li> </ul> | <ul> <li>Wear activity tracker for 7 days prior to starting the study intervention (use encouraged but not required throughout the study intervention period)</li> <li>Complete the Sleep Diary for 7 days prior to starting the study intervention</li> </ul> | <ul> <li>Wear activity tracker (and other study devices, if applicable, as specified in your Sub-Study Consent Form); use encouraged beginning at week 2</li> <li>Safety assessment</li> <li>Provide details about how you are completing your sub-study intervention(s)</li> <li>Wear activity tracker (and other study devices, if applicable, as specified in your Sub-Study Consent Form) and complete the Sleep Diary for the last 7 days before the final in-person visit</li> </ul> |

<sup>\*</sup>Stool samples will be collected after the visit with a home stool sample collection kit

<sup>\*\*</sup>Refer to your Sub-Study Consent Form for additional activities



Duke Clinical Research Institute (DCRI) / Protocol Number Pro00112484 / RECOVER-SLEEP


| Final In-Person Visit** | 1 Week Before the Final Phone Call** | Final Phone Call (end of study) ** |
|---|---|---|
| Clinic Visit | At-Home Activities (Phone and Internet-<br>Based) | At-Home Activities (Phone and Internet-Based) |
| <del>1</del> | | |
| Questionnaires and brain quizzes | Wear activity tracker for 7 days before the | Questionnaires |
| Review medications | final phone call | Safety assessment |
| Sleep history | | |
| Measure weight | | |
| <ul><li>Blood collection</li><li>Stool Sample*</li></ul> | | |
| Safety assessment | | |
| <ul> <li>Provide details about how you are completing the<br/>study intervention(s)</li> </ul> | | |
| <ul> <li>Return study materials (study drugs, study devices,<br/>etc.), as applicable</li> </ul> | | |

<sup>\*</sup>Stool samples will be collected after the visit with a home stool sample collection kit

<sup>\*\*</sup> Refer to your Sub-Study Consent Form for additional activities

SD\_ICF\_V3.0\_ 

#### What if I decide to stop participating before the study is over?

You can stop participating in this study at any time. If possible, we would like you to stay in the study until it is over because your information and experiences are valuable to this research. Even if you stop the study intervention early, such as stopping the study drug, we may ask that you continue to complete the study visits, if and when possible.

If you are thinking about stopping your participation, please let your study doctor know as soon as possible. Your study doctor can talk to you about options that might work for you to stay in the study, though you may continue to stop your participation if you so choose.

We will tell you if we learn anything new that might affect your decision about whether to continue participating in the study. If we lose contact with you, you will be automatically withdrawn from the study, and no further information will be collected from your medical record.

Your participation in the study may be stopped by your study doctor at any time without your consent. The study doctor may stop the study and end your participation at any time for any reason in order to ensure your safety. Some of the possible reasons include:

- Failure to follow study instructions.
- Continuing could be harmful to you.
- Termination of the study.
- Other unanticipated circumstances.

If your participation is stopped by your study doctor without your consent, you will be notified of the decision and reasoning.

#### **HOW WILL YOU PROTECT MY PRIVACY?**

In all research, there is a possible risk of the loss of confidentiality. We will make every effort to keep your personal and health information secure, but absolute confidentiality cannot be guaranteed.

To help us protect your privacy, this study is covered by a Certificate of Confidentiality from the National Institutes of Health (NIH) and the U.S. Department of Health and Human Services. This means that the study team cannot share any information that could identify you with anyone who is not involved in the research except for specific situations, such as when it is required by law to report child or elder abuse, some communicable diseases, and threats to harm yourself or others. The study team cannot be forced to share information that could identify you for use as evidence in any court of law or legal processes unless you give your permission.



Duke Clinical Research Institute (DCRI) / Protocol Number Pro00112484 / RECOVER-SLEEP


Your information that is protected by the Certificate of Confidentiality may still be shared or used when the information:

- 1. Is disclosed to people connected with the research. For example, the information may be used internally by the NIH for program evaluation.
- 2. Is required to be disclosed by federal, state, or local laws. For example, when information must be disclosed to meet the legal requirements of the U.S. Food and Drug Administration (FDA).
- 3. Is necessary for your medical treatment and you have given your permission for the information to be shared.
- 4. Is used for other research that is allowed by federal regulations.
- 5. Is shared with your permission. For example, if an insurance or healthcare provider gets your written consent for us to disclose the research information.

## By signing and dating this consent form, you consent to your information being used as described above.

You should understand that a Certificate of Confidentiality does not prevent you or a loved one from voluntarily releasing information about yourself or your involvement in this research. If you want your research information to be released to an insurer, medical care provider, or any other person not connected with the research, you must give your permission for the researchers to release it. This means that you and your loved ones must also actively protect your own privacy.

Finally, you should understand that the study doctor is not prevented from taking steps to prevent serious harm to yourself or others, including reporting to authorities.

#### **Receiving Information from Your Medical Record**

We may review your medical record while you are in the study. Your medical record may include information about visits to your study site, the hospital, or emergency room during the study. We may also collect information about medicines, lab results from blood or urine tests, and other information that may be useful to the study. Reviewing your medical record will help us understand your health status while you are participating in the study.

#### **ALTERNATIVES**

#### What other choices are there?

Your other choice is not to participate. You can continue to get your usual healthcare whether or not you participate in the study.



Duke Clinical Research Institute (DCRI) / Protocol Number Pro00112484 / RECOVER-SLEEP


Currently, no FDA-approved medicines or interventions are available to treat Long COVID. However, other options may be available to you if you choose not to participate in this study. Talk to the study doctor or your healthcare provider about these other options. The study doctor will discuss with you the major risks and benefits of usual care and alternative options.

#### **RESULTS AND STUDY PROGRESS**

#### Will I be told the results of the research?

We will summarize what we have learned when the final study results become available. We will share the summary of results on the study website. However, we may contact you by email, letter, newsletters, or other updates related to the study prior to the final study results.

A description of this clinical trial will be available on http://www.clinicaltrials.gov, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

The research summaries or articles published about the study will not include any information that could identify you.

#### POSSIBLE RISKS AND DISCOMFORTS

A team of health experts called the Data and Safety Monitoring Board, chosen by the NIH, will regularly monitor the safety of study participants and the progress of the study overall.

Any intervention may have associated risks. Because of this, it is important to notify the study team of any new or worsening symptoms you may experience during or after using the study interventions. There may be unknown risks from participation. For information about the risks of the study interventions for each sub-study, refer to the Sub-Study Consent Form.

Below are some possible, known risks about the study activities. There is also the risk of loss of confidentiality. Every effort will be made to protect your information, as described throughout this consent form. There may also be risks from participation that we do not know about yet. Refer to your Sub-Study Consent Form regarding risks about the sub-study interventions and sub-study activities.

#### Risks Associated with Terms of Use

As part of this research, you may be required to use one or more of the following: a phone or web app/ site, an electronic study diary (eDiary), or a device that tracks information about you. While using these, information about you may be collected and shared with the researchers or



Duke Clinical Research Institute (DCRI) / Protocol Number Pro00112484 / RECOVER-SLEEP


people outside of the study. This data might include personal health information, location, call logs, text message history, web browsing history, or social media use. A complete description of the data collection and sharing for an app, electronic study diary (eDiary), or device can commonly be found in the Terms of Use, End User License Agreement, or Privacy Policy associated with the device. If you would like to read these documents, request a copy or instructions about how to access this information from the study doctor.

While the Terms of Use, End User License Agreement, or Privacy Policy may include statements limiting your rights if you are harmed as a result of your use of the app, electronic study diary (eDiary), or device in this study, you do not release the study doctor, sponsor, study site, or agents for responsibilities from mistakes. You also do not waive any of your rights as a research participant.

#### Risks Associated with Home Sleep Apnea Testing (HSAT)

Risks associated with home sleep testing include skin irritation, where sensors are taped to the skin, and temporary disturbance of sleep.

#### **Risks Associated with Blood Draws**

The risks of getting your blood drawn include bleeding at the puncture site, bruising, and pain. Bleeding and bruising occur in a very small number of people who have their blood drawn. A very short period of pain from the needle stick occurs in most people. Some people may become dizzy, lightheaded, or feel faint. On rare occasions, infection of the area where the blood was drawn may occur.



#### Risks Associated with Tests to Measure Memory and Thinking Abilities ("Brain Quizzes")

Brain Quizzes may cause frustration, tiredness, or headaches during and/or after completion.

#### **Risks Associated with Nasal Swabs**

The risks of nasal swabs include possible discomfort, mild irritation, mild local pain, and minor bleeding.

#### Risks Associated with Activity Tracking Wearable Study Devices

An activity tracking wearable study device (a Fitbit, or similar device) is a non-invasive device that records changes to your rest and activity patterns. The risks include possible irritation or discomfort where the study device is worn.

#### Risks Associated with Pregnancy While Participating

If you could become pregnant (you have not had a hysterectomy and/or both tubes and/or both ovaries removed and/or you are not postmenopausal and over the age of 45) and you have a sexual partner who is able to have children (has not had a vasectomy with a negative post-surgery semen analysis), you must avoid becoming pregnant during the study and for at least 7 days after finishing the study intervention. Avoiding pregnancy is important due to potential side effects of the study drugs. There may be unknown risks to a pregnancy, embryo, or fetus if you become pregnant. The study team can tell you about effective methods of birth control.

However, because no birth control method is 100% effective, except abstinence, you should notify your study doctor immediately if you think there is any chance you could be pregnant, even if you have had a recent negative pregnancy test. If you become pregnant, we may want to review your medical history before and after you give birth. The study team will ask pregnant participants to complete a pregnancy-specific consent form in order to follow the pregnancy to its outcome.

#### **Future Contact**

We may contact you to ask if you are interested in participating in additional research related to the RECOVER Initiative. The additional follow-up calls, visits, and/or participation in additional research are optional and are not included as part of this consent form. You will be asked to sign a separate consent form if you agree to participate in additional research.

#### **BIOREPOSITORY: RESEARCH USE OF DATA AND BIOSPECIMENS**



A biospecimen is a sample such as urine or blood collected from the body for tests. With your permission, the biospecimens collected during this study—blood, and stool (poop), —will be sent to a storage place called the RECOVER Research Biorepository at Mayo Clinic in Rochester, Minnesota. These samples will be used for research on COVID and the long-term effects of COVID, but they may also be used for research on other health problems.

#### Why are biospecimens needed?

Biospecimens can provide valuable information to researchers. For example, blood contains substances like hormones, antibodies, and other things that can be measured. New substances are still being discovered, and methods for measuring these substances are being developed all the time. Tests to measure the amount or presence of a substance are used by doctors to assess health.



Duke Clinical Research Institute (DCRI) / Protocol Number Pro00112484 / RECOVER-SLEEP


Some substances found in biospecimens are called "biomarkers." Biomarkers can be measured and may provide important information about Long COVID. Blood sugar level is an example of a biomarker for diabetes. Biomarkers may also predict how a patient will respond to a treatment.

#### How will my biospecimens be used for research?

For this study, biospecimens will be used to try to understand how the study intervention may impact the immune system (body's defense against infection). We will also look for evidence that the virus that causes COVID-19 or that other infectious agents can be identified in the biospecimens. The collection of these biospecimens is required as part of this study.

We would also like to make your data and biospecimens available for future research. The research may be about similar diseases or conditions related to this study. However, research could also be about unrelated diseases, conditions, or other types of research. These studies may be done by researchers at this study site or other institutions, including commercial entities.

Although you will not receive any direct benefits, sharing your data and biospecimens with the RECOVER Research Biorepository may:

- Contribute to research that could help others in the future and improve medical care and public health
- Help researchers make important discoveries about medical conditions and possible therapies
- Improve our understanding of how study drugs and other interventions may work to reduce Long COVID symptoms
- Increase the possibility of developing new interventions and treatments related to Long COVID
- Enhance our understanding of how and why Long COVID affects people differently

#### Will my biospecimens be used for genetic testing?

The use of your samples for genetic testing is optional. At the end of this consent form, you will have the chance to tell us whether or not you want to allow researchers to use the samples we collect for genetic testing. Genetic testing looks at your DNA, the material that makes up your genes. Genes are the part of cells that tell our bodies how to grow and function, and they are passed from parent to child. Researchers may also perform a whole genome analysis on your DNA samples. Usually, researchers study just a few areas of your genetic code that are linked to a disease or condition. In whole genome studies, all or most of your genes are analyzed and used to study links to Long COVID. Genetic tests can determine if a person or groups of people are more likely to have certain genetic diseases or conditions.



Duke Clinical Research Institute (DCRI) / Protocol Number Pro00112484 / RECOVER-SLEEP


#### Will researchers be able to identify me based on my data and biospecimens?



We will do our best to protect your data and biospecimens during storage and when they are shared. However, there remains a possibility that someone could identify you. There is also the possibility that unauthorized people might access your data and biospecimens. In either case, we cannot reduce the risk to zero.

To protect your privacy, your name and identifying information will be removed from any data and biospecimens you provide before they are shared with other researchers. Your deidentified data and biospecimens may be shared with researchers around the world. However, the decision to share your data is controlled by the National Institutes of Health (NIH). To get your data and biospecimens, future researchers must seek approval from the NIH. The data and biospecimens submitted to a storage place or shared for research use will not include any information that can personally identify you, and researchers cannot easily link your identifying information to the data and biospecimens.

Genetic Information Nondiscrimination Act. Your data and biospecimens from this study are also protected by a federal law in the United States called the Genetic Information Nondiscrimination Act (GINA), which prevents health insurers from using genetic information to determine the cost of health insurance and prevents certain genetic discrimination. GINA does not protect against genetic discrimination by companies that sell life insurance, disability insurance, or long-term care insurance. GINA does not protect you against discrimination based on a genetic disease or condition that is already diagnosed.

#### Will I need to give additional permission for researchers to use my data?

No. The research use or sharing of your data and biospecimens can be done without getting additional permission from you. However, all future research studies will be approved by an independent scientific committee or ethics board.

#### Will I be paid for any future use of my data and biospecimens?

No. You will not be paid for any future use of your data or biospecimens. Your data and biospecimens will not be sold, but the use of your information or samples may lead to new tests, drugs, devices, or other products or services with commercial value. These products or services could be patented or licensed. There are no plans to provide any payment to you should this occur.



Duke Clinical Research Institute (DCRI) / Protocol Number Pro00112484 / RECOVER-SLEEP


#### How long will my data and biospecimens be stored for future use?

Your data will be stored indefinitely. Your biospecimens from this study will be kept until they are used up.

#### Will I get any results back from future research use of my data and biospecimens?

No. You should not expect to receive results from any future research that may use your data and biospecimens.

#### What if I change my mind about future use of my data and biospecimens?

Participating in this study means you agree to share your data and biospecimens. You can change your mind later, but researchers might still use your data and biospecimens if they have already been shared. If you do not want your data and biospecimens used for other research projects, you should not participate in this study.

If you decide that you do not want us to use or share your data and biospecimens, you can contact your study site to request they destroy any remaining samples. Please see the contact information at the beginning of this consent form. You will be notified of compliance with such a request, and supporting materials will be maintained for tracking.

If we are not able to link your samples back to you because they have already been deidentified, we will not be able to locate the samples to destroy them. In addition, if the data are needed to preserve the integrity of the study database for regulatory purposes, we will not be able to remove individual data until the regulatory processes are completed. We will also not be able to destroy any samples that have already been used or shared.

#### **PAYMENT AND COSTS**

#### Will I be paid for being in this study?

«Compensation»

If you participate in a sub-study, you may receive up to \$700 to cover study-related costs such as parking, and for your time and effort to complete the visits. You will receive:

- \$250 after completing the randomization visit
- \$50 after completing the middle of study phone call
- \$350 after completing the final in-person visit
- \$50 after completing the final phone call

For Biorepository Samples, you may also receive up to \$300 for your stool samples (\$0 for the first sample, and \$300 for the second sample).

Duke Clinical Research Institute (DCRI) / Protocol Number Pro00112484 / RECOVER-SLEEP


#### Do I have to pay anything to be in this study?

No. There will be no charge to you or your health insurance provider for taking part in this study. All tests and the study interventions that are needed for this study that are not part of your usual medical care will be covered by the study. "Usual medical care" is the care you would receive whether or not you are part of this study. If you receive your usual medical care during the study, your health insurance provider will be billed for that care, as it is unrelated to the study.

## What should I do if I become ill or injured during the study?

If you become ill or are injured while you are in the study, get the medical care that you need right away. You should inform the healthcare provider treating you that you are participating in this study. If you tell the study team that you think you have been injured, they will help you get the care you need.

However, there is no commitment by **the study site**, your healthcare providers, study drug or study device providers, study doctors, Duke University (Duke Clinical Research Institute), or the NIH to provide monetary compensation or free medical care to you in the event of a study-related injury. The Sponsor has no plans to pay for the cost of any additional care beyond what is provided as part of the study.

By signing this document, you will not lose any of your legal rights or release anyone involved in the research from responsibility for possible mistakes.

#### **USE OF PROTECTED HEALTH INFORMATION FOR RESEARCH**

#### What is Protected Health Information (PHI)?

The PHI collected for this research study includes your name, address, phone number, email address, date of birth, Social Security number, and health information.



#### Will my PHI remain private?

We will make every effort to keep your PHI safe. We will store records in a locked cabinet or office or on a password-protected computer. We will assign your study information a code and keep it separately from your personal record. Your identity and your PHI will not be shared unless it is required to protect your safety, the safety of others, or if you give us permission to share it.



Duke Clinical Research Institute (DCRI) / Protocol Number Pro00112484 / RECOVER-SLEEP


#### Who will have access to or receive my PHI?

Your PHI may be given to others only if needed for reasons like determining the results of the study, making sure the study is being done correctly, and providing required reports.

Your medical and research records may be accessed by:

- Your study doctor and other study team members.
- The Sponsor (DCRI) and its representatives (including its affiliated companies that help carry out the research).
- People, or organizations providing services for, or collaborating with, the Sponsor.
- Other researchers, including researchers involved in the study at study sites other than the one where you are participating in the study.
- Any organization that obtains all or part of the Sponsor's business or rights to the product under study.
- Government or regulatory authorities, such as the FDA, including those located in other countries.
- Advarra Institutional Review Board, an independent committee established to oversee the study and help protect the rights of research participants.
- A team of health experts called the Data and Safety Monitoring Board, chosen by the NIH, who will regularly monitor the safety of study participants and the progress of the study overall.

#### In addition:

• If we cannot reach you during the study period to confirm your health status, we may search for you or delegate a search for you using publicly available data to check on your well-being and health status.

Those who receive your information for the purpose of conducting the study may share it without your permission. Federal privacy rules may not apply to these groups; however, they have their own rules and codes to assure that all efforts, within reason, will be made to keep your PHI private.

#### How long will you keep my PHI?

We will keep your permission to use and share your PHI unless you take it back sooner. In California and any other state that requires an expiration date, the Authorization will expire 50 years after you sign and date this authorization document.





Duke Clinical Research Institute (DCRI) / Protocol Number Pro00112484 / RECOVER-SLEEP


You may take back your permission to use and share your PHI at any time by writing to the study doctor at the address listed on page 1 of this consent form. If you do this, you will not be able to stay in this study. No new PHI will be collected after your written request is received. However, PHI that has already been collected may still be used and given to others as described in this authorization form.

#### What about my medical record?

Information about your participation in this research will be in your medical record. Other than you, only people who have access to your medical record (like your study doctor and the study team) will be able to see this part of your medical record. The study team may send copies of parts of your medical record to the Duke Clinical Research Institute (DCRI) to monitor the study. Monitoring means DCRI staff will review study records, including your signed consent, to make sure that your information was entered correctly in the study records.

Like all your other information, we will keep this data as safe and secure as possible.

During the study, you will not be able to access your health data in the study records to make sure the study results are accurate. You will be able to access your study health data when the study is over.

#### What happens if I do not want to share my PHI with you?

If you decide not to sign this authorization form, you will not be able to take part in the study. If you take back your permission for us to use your PHI, you will not be able to continue in this study.

#### How can I learn more about my legal rights while participating in this study?

After declaring COVID-19 to be a public health emergency, the US Department of Health and Human Services issued a public health declaration called the Public Readiness and Emergency Preparedness Act Declaration for Countermeasures Against COVID-19 (PREP). Since being issued in March 2020, PREP has limited the legal rights of a subject participating in a COVID-19 clinical study that uses a drug, device or vaccine designed to treat, diagnose, cure or prevent COVID-19.

The ending of the public health emergency on May 11, 2023 does not automatically terminate PREP coverage for activities related to COVID-19. Whether PREP can continue to limit the legal rights of subjects participating in a COVID-19 clinical study after the public health emergency ends depends on a number of complex factors that can be subject to change. If PREP limitations on subjects' legal rights apply to the study drug(s) and study device(s), subjects using



 $SD\_ICF\_V3.0\_$ 

Duke Clinical Research Institute (DCRI) / Protocol Number Pro00112484 / RECOVER-SLEEP


the study drug(s) and study device(s) in the study may have limits on their right to sue the manufacturers, the study sponsor, healthcare providers and others for significant injuries and adverse reactions.

## **OPTIONAL: SAMPLE COLLECTION FOR GENETIC TESTING**

| | tic testing. By initialing below, you confirm you have been told that e study without providing samples for genetic testing. |
|---|---|
| Initials | <b>Yes,</b> I give study team permission to collect samples for future unspecified genetic testing. |
| Initials | <b>No,</b> I do not give study team permission to collect samples for future unspecified genetic testing. |

Please initial the appropriate line below to let us know whether or not you want to allow your

 $SD\_ICF\_V3.0\_$ 

Duke Clinical Research Institute (DCRI) / Protocol Number Pro00112484 / RECOVER-SLEEP


## STATEMENT OF AUTHORIZATION

I have read this authorization form, its contents were explained, and my questions have been answered. I voluntarily agree to allow the study team to collect, use, and share my personal and health information as specified in this authorization form. I will receive a signed and dated copy of this authorization form for my records. I understand that I am not giving up any of my legal rights by signing this form.

| Participant: | |
|---|---|
| Print name: | |
| Signature: | |
| Date: | Time: |
| The study part<br>has been read<br>by a member o | IATURE FOR PARTICIPANTS WHO CANNOT READ cicipant has indicated that he/she is unable to read. This Authorization document to the participant by a member of the study team, discussed with the participant of the study team, and the participant has been given an opportunity to ask ne study team. |
| Print name: | |
| Signature: | |
| Date: | Time: |

SD\_ICF\_V3.0\_ 

#### WHOM TO CONTACT ABOUT THIS STUDY

During the study, if you experience any medical problems, suffer a research-related injury, or have questions, concerns or complaints about the study such as:

- Whom to contact in the case of a research-related injury or illness;
- Payment or compensation for being in the study, if any;
- Your responsibilities as a research participant;
- Eligibility to participate in the study;
- The study doctor's or study site's decision to withdraw you from participation;
- Results of tests and/or procedures;

## <u>Please contact the study doctor at the telephone number listed on the first page of this consent document.</u>

If you seek emergency care, or hospitalization is required, alert the treating physician that you are participating in this research study.

An institutional review board (IRB) is an independent committee established to help protect the rights of research participants. If you have any questions about your rights as a research participant, contact:

By mail:

Study Subject Adviser Advarra IRB 6100 Merriweather Dr., Suite 600 Columbia, MD 21044

• or call **toll free**: 877-992-4724

• or by **email**: adviser@advarra.comadviser@advarra.com

Please reference the following number when contacting the Study Subject Adviser: <u>Pro00073133.</u>



Duke Clinical Research Institute (DCRI) / Protocol Number Pro00112484 / RECOVER-SLEEP


#### STATEMENT OF CONSENT

A copy of this consent form will be given to you. The purpose of this study, the procedures to be followed, and the risks and benefits have been explained to me. I have been allowed to ask questions, and my questions have been answered to my satisfaction. I have been told who to contact if I have questions, to discuss problems, concerns, or suggestions related to the research, or to get information about the research. I have read this consent form and agree to be in this study, with the understanding that I may withdraw at any time. I have been told that I will be given a signed and dated copy of this consent form.

| Participant: | |
|--------------|------------------|
| Print name: | |
| Signature: | |
| Date: | Time: |
| Person Who O | btained Consent: |
| Print name: | |
| Signature: | |
| Date: | Time: |



 $SD\_ICF\_V3.0\_$ 

Duke Clinical Research Institute (DCRI) / Protocol Number Pro00112484 / RECOVER-SLEEP


#### WITNESS SIGNATURE FOR PARTICIPANTS WHO CANNOT READ, IF APPLICABLE

The study participant has indicated that he/she is unable to read. The consent document has been read to the participant by a member of the study team, discussed with the participant by a member of the study team, and the participant has been given an opportunity to ask questions of the study team.

| Print name: | |
|-------------|-------|
| Signature: | |
| Date: | Time: |